CLINICAL TRIAL: NCT03777826
Title: An Open-label, Explorative, Post Launch, Multicenter, Multi-country Intervention Study of PKU Synergy (an Amino-acid Mixture) to Evaluate Change in Nutrient Intake in PKU Subjects With an Increased Phe-tolerance/Intake
Brief Title: Effects of Synergy on Nutrient Intake and Acceptability in Phenylketonuria (PKU)
Acronym: ESSENTIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPR16TA09791
Record Dates: First submitted 2018-11-19; First posted 2018-12-17 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open label (1 arm) (Other): Open label use of study product (post-marketing): PKU Synergy
  Interventions: Other: PKU Synergy

INTERVENTIONS:
Other: PKU Synergy — PKU Synergy is a citrus flavored, powdered amino-acid mixture (containing traces of Phe, 4,3mg per portion; and 20 gr. Protein Equivalent (PE)) with a tailored amino acid and micronutrient profile adapted for the special requirements of HPA/PKU (Hyperphenylalaninemia/Phenylketonuria) subjects over 10 years of age with an increased Phenylalanine-(Phe) tolerance/intake.

SUMMARY:
Phenylketonuria (PKU) is a rare inherited metabolic disorder, where subjects are born with a genetic deficiency in the phenylalanine hydroxylase enzyme (PAH), which leaves them unable to convert Phenylalanine (Phe) into Tyrosine (Tyr). Patients with mild PKU or partly responsive to the drug synthetic tetrahydrobiopterin (BH4) (Kuvan®) can change to a more relaxed diet. However due to difficulty to adapt their diet, these patients are at risk of an imbalanced nutritional status and an insufficient intake of specific micronutrients, essential amino acids and DHA (Docosahexaenoic acid). The study product is designed to improve the nutritional status of the patients.

The study investigates if the nutritional status is indeed improved following 24 week use of the study product, and also the study aims to evaluate product acceptability.

ELIGIBILITY:
Inclusion criteria:

1. PKU subjects identified by newborn screening and started low-Phe diet before 3 months of age
2. PKU subjects (with or without current AAM use) with an increased Phe-tolerance/intake due to:

   * Mild PKU phenotype
   * BH4 treatment
3. If treated with BH4, PKU subjects should be on a stable BH4 treatment for at least 26 consecutive weeks up to start test product intake
4. Age≥12 years
5. If subjects (irrespective whether BH4 users or mild PKU) use amino-acid mixture(s; AAM), then a maximum of 25 Protein Equivalents (PE) derived from the AAM per day applies and usage on a daily basis for at least 26 consecutive weeks up to Visit 1
6. If subjects (irrespective whether BH4 users or mild PKU) use AAMs they should be capable and willing to substitute their current AAM(s; maximum of 25 PE per day) with one portion of the test product per day
7. If subjects (irrespective whether BH4 users or mild PKU) use omega-3, antioxidant, and/or vitamin supplements, to stop usage of the supplements and be able and willing to substitute with the test product
8. Willing and able to comply with study procedures
9. Willing and able to provide informed consent (and assent in case of minors if required by local law/regulations)
10. For women of childbearing potential: not to have the intention to become pregnant during the study

Exclusion Criteria:

1. For women: Currently pregnant or lactating
2. Current or prior use of the test product within six weeks prior to entry into the study
3. Concurrent conditions (including renal failure and severe hepatic failure) and medication that could interfere with participation, outcome parameters or safety (as determined by Investigator)
4. Psychotropic medication (i.e. medication affecting the nervous system) and inotropic medication
5. Any condition creating high risk of poor compliance with study
6. Participation in any other studies involving investigational or marketed products concomitantly or within six weeks prior to entry into the study. Except for studies related to Kuvan® (synthetic tetrahydrobiopterin (BH4)) without diagnostic, therapeutic or experimental intervention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Nutrient intake | 24 weeks
  Change in nutrient intake after 24 weeks by analysis of 3 day diet diary. Nutrients (energy, micronutrients, essential amino acids and DHA) in [(m)/(micro)gram/day] or [mg/day or mg/kg/day]
Product acceptability | 24 weeks
  Product acceptability questionnaire [category/score] [0-10] and [0-5]

SECONDARY OUTCOMES:
Compliance | 24 weeks
  Compliance (product consumption) using daily product intake diary [number of products used per week; per sachet of 33g]
Phenylalanine (Phe) levels | 24 weeks
  Dried bloodspot Phenylalanine (Phe) levels [µmol/L]
Blood chemistry: nutritional status | 24 weeks
  Blood chemistry: levels measured in blood: Full Fatty acid profile [For each FA Erythrocyte Membranes level (%FA)], full Amino acid profile [µmol/L], Vitamin B12 [pM], Vitamin D [ng/ml /nmol/L]; Folic acid [nM]; Selenium [µM]; Iodine [µg/L/ ng/mL]; Calcium [mg/dL]; Zinc [µmol/L]; Iron [µg/L] analyzed in blood samples by central laboratories
Anthropometrics: weight | 24 weeks
  Anthropometrics: Weight [kg]
Anthropometrics: height | 24 weeks
  Anthropometrics: Height [cm or m]
Anthropometrics: BMI | 24 weeks
  Anthropometrics: BMI [kg/m2], calculated from weight/height

OTHER OUTCOMES:
Safety Parameters (Incidence, frequency, seriousness, severity and relatedness of (Serious) Adverse Events) | 24 weeks
  Incidence, frequency, seriousness, severity and relatedness of (Serious) Adverse Events
Tolerance (Standard gastrointestinal questionnaire reporting) | 24 weeks
  Tolerance: Standard gastrointestinal questionnaire reporting of diarrhea constipation, abdominal distension, nausea, vomiting, burping, flatulence, regurgitation, and colic/cramps (0, 1, 12 and 24 weeks) [absent, mild, moderate, severe]
Subject characteristics | week 0
  * Age [years]
  * Sex [male/female]
  * Country [Germany/Netherlands]
Phe tolerance level and/or range | week 0
  [mg Phe/day]
PKU phenotype | week 0
  Recording of PKU (Phenylketonuria) genotype from medical history [hyperphenylalaninemia (HPA) or mild/moderate/classic PKU]

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (2):
  - University hospital Leipzig, Leipzig
  - University hospital Münster, Münster
- University Medical Center Groningen (UMCG), Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No